CLINICAL TRIAL: NCT04502277
Title: Comparative,Randomized,Single-dose,2-way Crossover Bioavailability Study of 40mgm/ml 35 ml Suspension and Pfizer (Diflucan®) 40 mg/ml 35 ml Fluconazole Suspension of Participants Under Fed Condition
Brief Title: Bioavailability of Flucanazole
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sutphin Drugs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Diflucan
Record Dates: First submitted 2020-07-31; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Candidiasis
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Flucanazole (Experimental): The Objective of This Study Was an Open-label, Randomized, 2-way Crossover to Compare the Single-dose Relative Bioavailability of Flucanazole 40mgm/ml 35 ml Suspension and to measure AUC at 0, 1 , 4 , 8, 12, 16 , 20 and 24 hours Under Fed Condition
  Interventions: Drug: Fluconazole Powder
- Diflucan (Active Comparator): The Objective of This Study Was an Open-label, Randomized, 2-way Crossover to Compare the Single-dose Relative Bioavailability of Diflucan 40mgm/ml 35 ml Suspension and to measure AUC at 0, 1 , 4 , 8, 12, 16 , 20 and 24 hours Under Fed Condition
  Interventions: Drug: Fluconazole Powder

INTERVENTIONS:
Drug: Fluconazole Powder — The Objective of This Study Was an Open-label, Randomized, 2-way Crossover to Compare the Single-dose Relative Bioavailability of Diflucan 40mgm/ml 35 ml Suspension and to measure AUC at 0, 1 , 4 , 8, 12, 16 , 20 and 24 hours Under Fed Condition

SUMMARY:
The Objective of This Study Was an Open-label, Randomized, 2-way Crossover to Compare the Single-dose Relative Bioavailability of Flucanazole 40mgm/ml 35 ml Suspension and Pfizer (Diflucan®) 40 mg/ml 35 ml Fluconazole Suspension Under Fed Condition

DETAILED DESCRIPTION:
The study is to be conducted as an open-label, randomized, single-dose, 2-way crossover, relative bio availability study performed on 200 healthy adult volunteers. A total 200 subjects will be assessed for AUC for 72 hours after administration of flucanazole suspension

ELIGIBILITY:
Inclusion Criteria Male and females between the ages of 18 and 35 years

* Healthy Individual
* Able to swallow

Exclusion Criteria:

* History or presence of significant:

  * cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.

In addition, history or presence of:

alcoholism or drug abuse within the past year; hypersensitivity or idiosyncratic reaction to fluconazole or other azoles. Subjects who have used any drugs or other substances known to be strong inhibitors of CYP (cytochrome P450) enzymes within 10 days prior to first dose.

Subjects who have used any drugs or other substances known to be strong inducers of CYP (cytochrome P450) enzymes within 30 days prior to first dose.

Subjects who have been anormal diet during the 30 days prior to the first dosing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Bio availability | 24 hours
  To measure the AUC at 0, 1 , 4 , 8, 12, 16 , 20 and 24 hours after a single dose administration of Under Fed Condition

CONTACTS AND LOCATIONS:
Locations (2):
- Sutphin Drugs, Jamaica, New York, United States
- Lifein Multi-Specialty Hospital, Navsari, Gujarat, India

IPD SHARING:
Plan to Share IPD: No